CLINICAL TRIAL: NCT07267364
Title: Comparison of Pelvic Floor Muscle Training and Dynamic Neuromuscular Stabilization Exercises in Pediatric Patients Diagnosed With Voiding Dysfunction: A Randomized Controlled Trial
Brief Title: Comparison of Pelvic Floor Muscle Training and Dynamic Neuromuscular Stabilization Exercises in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Saliha Özer, Physıcal Therapy and Rehabilitation, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23743.R1
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Urology; Pediatric Disorder
MeSH Terms: interventions — pentalenolactone F methyl ester

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Education group (PFME) (Active Comparator): Children diagnosed with dysfunctional voiding will receive pelvic floor training using superficial video visuals, and pelvic muscle strength and endurance will be increased with EMG and biofeedback. Exercises will be administered three days a week for approximately eight weeks. They will be assessed before and after treatment with the Voiding Disorders Symptom Score (VDSS), the Children's Depression Scale, the Quality of Life for Children with Urinary Incontinence (QOLS), the Bladder and Bowel Dysfunction Scale (BDS), the Stool Scale, and the Children's Body Image Scale.
  Interventions: Behavioral: PFME
- PFME+DNS group (Active Comparator): In addition to PFME, an exercise model that begins with Dynamic Neuromuscular Stabilization (DNS) spine stabilization and addresses muscle synergies will be applied for approximately 8 weeks. hey will be assessed before and after treatment with the Voiding Disorders Symptom Score (VDSS), the Children's Depression Scale, the Quality of Life for Children with Urinary Incontinence (QOLS), the Bladder and Bowel Dysfunction Scale (BDS), the Stool Scale, and the Children's Body Image Scale.
  Interventions: Behavioral: PFME

INTERVENTIONS:
Behavioral: PFME — During PFME, children are taught about the pelvic floor using video visuals and their awareness of the pelvic floor muscles is increased. They are then instructed on how to contract and relax their muscles to control urination. DNS exercises, on the other hand, is an exercise model that begins with spinal stabilization and focuses on muscle synergies. Participants in the study will be assessed twice: at the beginning and end of treatment, using the Voiding Disorders Symptom Score (VDSS), the Quality of Life for Children with Urinary Incontinence (QOLQ), the Bladder and Bowel Dysfunction Scale (BBS), the Bristol Stool Scale, and the Children's Body Image Scale.
  Other Names: PFME+DNS Exercise

SUMMARY:
Dysfunctional voiding (DY) is one of the most common conditions in children. Various treatments are available. Participants will be randomly assigned to either PTCE (Group I) or PTCE+DNS (Group II). PTCE is the gold standard and routinely administered in hospitals for children diagnosed with dysfunctional voiding who are referred by a urologist. The PTCE group serves as the control group, and treatment will be scheduled for a total of 10 weeks, two days a week. During PTCE, children receive instruction about the pelvic floor using video visuals and increase awareness of their pelvic floor muscles. They are then instructed on how to contract and relax their muscles to control urination. DNS training is an exercise model that begins with spinal stabilization and addresses muscle synergies. Patients included in the study will be evaluated twice, at the beginning and at the end of the treatment, with the Voiding Disorders Symptom Score (VODS), Quality of Life Scale for Children with Urinary Incontinence (QOLS), Bladder Bowel Dysfunction Scale (BDS), Bristol Stool Scale and Children's Body Image Scale.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with voiding dysfunction according to ICCS diagnostic criteria in a urology outpatient clinic,
* Being 5-18 years old,
* The child and their parent/guardian agree to participate in the study voluntarily and provide signed consent.

Exclusion Criteria:

* Organic pathologies such as urethral obstruction, ectopic ureter, spinal dysraphism, and diabetes
* Diagnosis of VUR or neurogenic bladder
* Cognitive and mental impairment
* Having spina bifida
* Being under 5 years of age
* Receiving treatment such as PTC training or electrical stimulation

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Voiding Disorders Symptom Scoring (VDSS) | baseline, post treatment (at 8 week)
  There are 13 questions about lower urinary tract symptoms and 1 question about quality of life. Regarding nocturnal enuresis, the frequency and severity of nocturnal enuresis are questioned. The total score ranges from 0 to 35 points, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Pediatric Quality of Life Questionnaire (PEDSQL) | baseline, post treatment (at 8 week)
  It consists of 23 items and four subsections. It covers physical health, emotional, social, and school functioning. Each item receives a raw score between 0 and 4. "0" = No problem, "1" = Almost no problem, "2" = Sometimes a problem, "3" = Usually a problem, and "4" = Almost always a problem. The resulting raw scores are rescored to range from 0 to 100 (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). A higher total score indicates a higher quality of life.
Children's Body Image Scale | baseline, post treatment (at 8 week)
  Body image will be measured using the Children's Body Image Scale. The scale has separate versions for boys and girls. The scale contains seven gender-specific images in anatomical positions. Each version includes seven male and seven female photos in the scale. Each photo represents a different BMI range. The images are ranked from A to G according to increasing BMI. Children will be asked to mark the image that best reflects their perceived body size and shape. The calculation will be made by subtracting the number equivalent to their actual BMI from the perceived number. The score range is from -6 to +6, with negative scores indicating a perception of self as smaller than they actually are, zero indicating a correct answer, and positive scores indicating a perception of self as overweight.
Depression Scale for Children | baseline, post treatment (at 8 week)
  Children's depression levels were assessed using the Children's Depression Scale, developed by Kovacs in 1981. The scale is applicable to children aged 6-17. Its validity and reliability in Turkish were demonstrated by Öy (1991). The scale consists of 27 items and has three different response options for each item. In our study, children were asked to think back over the past two weeks and select the sentence that best fits them. Each sentence set includes statements related to symptoms of childhood depression (e.g., sleep and appetite problems, dysphoria). Each sentence set can be scored between 0 and 2. Possible responses for each sentence set are "1. I sometimes feel sad," "2. I often feel sad," and "3. I always feel sad." The maximum score is 54. Higher scores indicate greater depression severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Konya, Konya
  - Hanife Dogan, Konya, Konya

IPD SHARING:
Plan to Share IPD: Undecided